CLINICAL TRIAL: NCT04407481
Title: PENGUIN: PErfusioN, OxyGen ConsUmptIon and ENergetics in ADPKD
Brief Title: PErfusioN, OxyGen ConsUmptIon and ENergetics in ADPKD (PENGUIN)
Acronym: PENGUIN
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0277
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Polycystic Kidney Disease, Adult; Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — During the study, we will collect blood and urine samples for assessment of kidney function and kidney injury markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults with autosomal dominant polycystic kidney disease: All participants will undergo DXA scan, PET/CT using 11-C acetate to measure renal oxygen consumption, hyperinsulinemic-euglycemic clamp to quantify insulin sensitivity, and renal clearance testing using iohexol and para-aminohippurate (PAH) to quantify glomerular filtration rate (GFR) and effective renal plasma flow (ERPF).
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 milligrams per milliliter (MG/ML); Radiation: PET/CT Scan
- Healthy Controls: Comparative data will be provided from healthy adults from an ongoing study with similar study design and methods (CROCODILE Study: Control of Renal Oxygen Consumption, Mitochondrial Dysfunction, and Insulin Resistance).

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: •- Sodium 4-amino hippurate (PAH) inj 20% 2g/10 milliliter (mL) • Para-aminohippurate • Aminohippuric acid
  Groups: Adults with autosomal dominant polycystic kidney disease
Drug: Iohexol Inj 300 milligrams per milliliter (MG/ML) — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300
  Groups: Adults with autosomal dominant polycystic kidney disease
Radiation: PET/CT Scan — Imaging used to visualize the kidneys and quantify renal metabolic activity
  Groups: Adults with autosomal dominant polycystic kidney disease

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common monogenic cause of end-stage kidney disease (ESKD). The disorder is characterized by development and continued growth of multiple cysts requiring renal replacement therapy in 50% of patients by age 60 years. However, ADPKD is also a complex metabolic disorder defined by insulin resistance (IR) and mitochondrial dysfunction which may be causally related to cyst expansion, kidney function decline and contribute to reduced life expectancy. Renal hypoxia, stemming from a potential metabolic mismatch between increased renal energy expenditure and impaired substrate utilization, is proposed as a novel unifying early pathway in the development and expansion of renal cysts in ADPKD. By examining the interplay between renal O2 consumption and energy utilization in young adults with and without ADPKD, the investigators hope to identify novel therapeutic targets to impede development of cyst expansion in future trials.

The investigators propose to address the specific aims in a cross-sectional study with 20 adults with ADPKD (50% female, ages 18-40 years). Comparative data will be provided from healthy adults from an ongoing study with similar study design and methods (CROCODILE Study: Control of Renal Oxygen Consumption, Mitochondrial Dysfunction, and Insulin Resistance). For this protocol, participants will complete a one day study visit at Children's Hospital Colorado. Patients will undergo a dual energy x-ray absorptiometry (DXA) to assess body composition, and a 11C-acetate positron emission tomography (PET/CT) scan to quantify renal O2 consumption. After the PET/CT, participants will undergo a hyperinsulinemic-euglycemic clamp while fasting to quantify insulin sensitivity. Glomerular Filtration Rate (GFR) and Effective Renal Plasma Flow (ERPF) will be measured by iohexol and PAH clearances during the hyperinsulinemic-euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Autosomal dominant polycystic kidney disease
* Age 18-40 years
* BMI >= 18.5 and <30 kg/m2
* Weight <350 lbs

Exclusion Criteria:

* Diabetes mellitus, based on previous diagnosis
* Albuminuria (≥30mg/g) or estimated glomerular filtration rate (eGFR) <75ml/min/1.73m2
* Pregnancy or nursing
* Anemia
* Allergy to shellfish or iodine
* Vaptan therapy (e.g. tolvaptan)
* Uncontrolled hypertension (average ≥140/90 mmHg)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The investigators propose to address the specific aims in a cross-sectional study with 20 adults with ADPKD (50% female, ages 18-40 years). Comparative data will be provided from healthy adults from an ongoing study with similar study design and methods.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Renal oxygen consumption | 30 minutes
  11-C Acetate PET/CT
Insulin Sensitivity | 4.5 hours
  Hyperinsulinemic-Euglycemic Clamp

SECONDARY OUTCOMES:
Mitochondrial Function | 5 minutes
  Blood draw for mitochondrial DNA copy number
Mitochondrial Function | 5 minutes
  Blood draw for untargeted metabolite assessment of the tricyclic acid (TCA) cycle
Mitochondrial Function | 5 minutes
  Blood draw for targeted assessment and quantification of glucose oxidation using an established metabolite panel
Mitochondrial Function | 5 minutes
  Blood draw for untargeted metabolite assessment of Free Fatty Acid (FFA) oxidation
Glomerular Filtration Rate (GFR) | 3 hours
  Iohexol Clearance Study
Effective Renal Plasma Flow (ERPF) | 2.5 hours
  PAH Clearance Study
Renin-Angiotensin-Aldosterone-System Activity | 5 minutes
  Blood draw for Plasma Renin levels
Renin-Angiotensin-Aldosterone-System Activity | 5 minutes
  Blood draw for Angiotensin II levels
Renin-Angiotensin-Aldosterone-System Activity | 5 minutes
  Blood draw for Copeptin levels
Kidney Injury Biomarkers | 5 minutes
  Chitinase-3-like protein 1 (YKL-40) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Neutrophil gelatinase-associated lipocalin (NGAL) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Kidney Injury Molecule 1 (KIM-1) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Interleukin-18 (IL-18) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for Tumor Necrosis Factor Receptor 1/2 (TNF-R 1/2) levels
Kidney Injury Biomarkers | 5 minutes
  Blood draw for monocyte chemoattractant protein-1 (MCP-1) levels

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bjornstad P, Richard G, Choi YJ, Nowak KL, Steele C, Chonchol MB, Nadeau KJ, Vigers T, Pyle L, Tommerdahl K, van Raalte DH, Hilkin A, Driscoll L, Birznieks C, Hopp K, Wang W, Edelstein C, Nelson RG, Gregory AV, Kline TL, Blondin D, Gitomer B. Kidney Energetics and Cyst Burden in Autosomal Dominant Polycystic Kidney Disease: A Pilot Study. Am J Kidney Dis. 2024 Sep;84(3):286-297.e1. doi: 10.1053/j.ajkd.2024.02.016. Epub 2024 Apr 15. PMID 38621633